CLINICAL TRIAL: NCT01138345
Title: The Effect of Chemotherapy on Aging in Older Women With Breast Cancer as Measured by Expression of p16INK4a
Brief Title: Biomarkers in Blood Samples From Older Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 0924; P30CA016086 (NIH); CDR0000674103 (Other: PDQ number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: cancer survivor; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Treatment w/Surgery: Breast Cancer survivors treated with surgery with or without radiation.
  Interventions: Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis; Other: medical chart review; Other: questionnaire administration
- Treatment w/endocrine therapy: Breast Cancer survivors treated with surgery with or without radiation plus endocrine therapy.
  Interventions: Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis; Other: medical chart review; Other: questionnaire administration
- Treatment w/ chemotherapy: Breast Cancer survivors treated with surgery with or without radiation and chemotherapy with or without endocrine therapy.
  Interventions: Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis; Other: medical chart review; Other: questionnaire administration

INTERVENTIONS:
Genetic: gene expression analysis — blood samples will be analyzed for the expression of the p16 gene.
Genetic: reverse transcriptase-polymerase chain reaction — perform reverse transcriptase-polymerase chain reaction on all blood samples.
Other: laboratory biomarker analysis — perform laboratory biomarker analysis on all blood samples
Other: medical chart review — perform medical chart review for all subjects
Other: questionnaire administration — each cohort will be given the same questionnaire

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers in blood samples from older women with stage I, stage II, or stage III breast cancer who have finished primary therapy or breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure and compare normalized p16^INK4a gene expression in women ≥ 65 years of age with stage I-III breast cancer who have completed primary therapy comprising surgery with or without radiotherapy followed by endocrine therapy (cohort 2) versus surgery with or without radiotherapy followed by chemotherapy and with or without endocrine therapy (cohort 3) .
* To measure and compare normalized p16^INK4a gene expression in women ≥ 65 years of age with stage I-III breast cancer who have completed primary therapy comprising surgery with or without radiotherapy (cohort 1) versus women treated in cohort 2.
* To compare normalized p16^INK4a gene expression between cohorts 1, 2, and 3 versus an age-matched contemporaneous control group of healthy volunteers accrued from a separate study (cohort 4).

Secondary

* To access functional status (ability to live independently at home and in the community), co-morbid medical conditions, cognition, psychological status, social functioning and support, medication review, nutritional status, and health-behavior status of these patients.

Tertiary (exploratory)

* To compare methodologies of p16 ^INK4a gene expression measurement in 50 patients in order to develop a batchable and analytically validated assay that eliminates the need for rapid sample processing.
* To explore any association between p16^INK4a expression and amount of vigorous physical activity, smoking habits, and/or weekly alcohol consumption.
* To explore any association between p16^INK4a expression and type of chemotherapy received, co-morbidities, concomitant medications, and/or tumor characteristics.
* To correlate p16^INK4a expression with scores from selected domains of the Geriatric Assessment (i.e., cognitive function, activities of daily living (ADL), and the instrumental ADL.

OUTLINE: Breast cancer survivors and healthy volunteers undergo blood collection for p16^INK4a gene expression analysis by Taqman RT-PCR.

Breast cancer survivors complete the Health Behavior and the Geriatric Assessment Questionnaires. They also complete a Timed Up and Go test to determine physical mobility.

Medical charts are reviewed to record information about diagnosis and treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage I-III disease
* Breast cancer survivors meeting 1 of the following criteria:

  * Prior surgery with or without (±) radiotherapy (RT) (cohort 1)
  * Prior surgery ± RT, followed by prior or concurrent hormonal (endocrine) therapy (cohort 2)

    * Must have received or be on endocrine therapy for ≥ 3 months
  * Prior surgery ± RT, followed by prior chemotherapy ± endocrine therapy (cohort 3)
* No recurrent disease
* No history of clonal bone marrow disorder (i.e., myelodysplastic or myeloproliferative disorder, acute or chronic leukemia)

PATIENT CHARACTERISTICS:

* Life expectancy > 12 months
* Absolute lymphocyte count > 500/μL
* No acute or active infection
* No other co-morbid illness that would impair ability to participate in the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior surgery with or without radiotherapy
* At least 3 months since prior chemotherapy (cohort 3)
* No concurrent radiotherapy, chemotherapy, or experimental therapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors age 50 and older who have completed their breast cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
p16INK4a expression between cohort 2 vs cohort 3 | 2 years
p16INK4a expression between cohort 1 vs cohort 2 | 2 years
p16INK4a expression between cohorts 1, 2, and 3 vs cohort 4 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States